CLINICAL TRIAL: NCT05267652
Title: Pragmatic Trial Examining Oxygenation Prior to Intubation
Acronym: PREOXI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Jonathan Casey, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211271
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Acute Respiratory Failure
Keywords: Critical illness; Emergency airway management; Tracheal intubation; Non-invasive ventilation; Facemask oxygen
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoxygenation with Non-Invasive Positive Pressure Ventilation Group (Active Comparator): Patients assigned to preoxygenation with non-invasive positive pressure ventilation will receive non-invasive mechanical ventilation via a tight-fitting mask from the initiation of preoxygenation until the initiation of laryngoscopy. Trial protocol will not dictate the brand or type of mechanical ventilator that will be used to deliver non-invasive ventilation.
  Interventions: Other: Preoxygenation with Non-Invasive Positive Pressure Ventilation
- Preoxygenation with Facemask Oxygen Group (Active Comparator): For patients randomized to preoxygenation with facemask oxygen, supplemental oxygen will be administered via a non-rebreather mask or bag-mask device without manual ventilation from the initiation of preoxygenation until induction. Trial protocol will not dictate the brand or type of facemask. The decision between use of a non-rebreather mask and use of a bag-mask device will be made by treating clinicians. The decision of whether to provide manual ventilation with a bag-mask device between induction and laryngoscopy will be made by treating clinicians.
  Interventions: Other: Facemask Oxygen

INTERVENTIONS:
Other: Preoxygenation with Non-Invasive Positive Pressure Ventilation — The delivery of oxygen and ventilation by non-invasive mechanical ventilation via a tight-fitting mask from the initiation of preoxygenation until the initiation of laryngoscopy. Trial protocol will not dictate the brand or type of mechanical ventilator that will be used to deliver non-invasive ventilation.
  Arms: Preoxygenation with Non-Invasive Positive Pressure Ventilation Group
Other: Facemask Oxygen — The delivery of supplemental oxygen via a non-rebreather mask or bag-mask device without manual ventilation from the initiation of preoxygenation until induction. Trial protocol will not dictate the brand or type of facemask. The decision between use of a non-rebreather mask and use of a bag-mask device will be made by treating clinicians. The decision of whether to provide manual ventilation with a bag-mask device between induction and laryngoscopy will be made by treating clinicians.
  Arms: Preoxygenation with Facemask Oxygen Group

SUMMARY:
Clinicians perform rapid sequence induction, laryngoscopy, and tracheal intubation for more than 5 million critically ill adults as a part of clinical care each year in the United States. One-in-ten emergency tracheal intubations is complicated by life-threatening hypoxemia. Administering supplemental oxygen prior to induction and intubation ("preoxygenation") decreases the risk of life-threatening hypoxemia. In current clinical practice, the most common methods for preoxygenation are non-invasive positive pressure ventilation and facemask oxygen. Prior trials comparing non-invasive positive pressure ventilation and facemask oxygen for preoxygenation have been small and have yielded conflicting results. A better understanding of the comparative effectiveness of these two common, standard-of-care approaches to preoxygenation could improve the care clinicians deliver and patient outcomes.

DETAILED DESCRIPTION:
BACKGROUND:

Clinicians frequently perform tracheal intubation of critically ill patients in the emergency department (ED) or intensive care unit (ICU). Complications of intubation, including hypoxemia and cardiovascular instability, occur in nearly half of intubations performed in these settings. Preventing complications during tracheal intubation is a key focus of clinical care and airway management research.

HYPOXEMIA DURING INTUBATION OF CRITICALLY ILL PATIENTS:

Life-threatening hypoxemia occurs in 1-in-10 cases of emergency tracheal intubation. Severe hypoxemia during intubation is associated with increased risk of cardiac arrest and death. Severe hypoxemia may be associated with worse outcomes in survivors. For example, neurologic recovery from traumatic brain injury may be worse after hypoxemia due to secondary ischemic insult.

ROLE OF PREOXYGENATION IN PREVENTING HYPOXEMIA DURING INTUBATION:

In current clinical practice, emergency tracheal intubation involves the nearly simultaneous administration of a sedative agent and a neuromuscular blocking agent to optimize the anatomic conditions for intubation. Following medication administration, patients rapidly become hypopneic and then apneic until invasive mechanical ventilation is initiated through the newly-placed endotracheal tube. The oxygen contained in the lungs at the time of neuromuscular blockade (i.e., the patient's functional residual capacity) is the reservoir of oxygen available to the patient's body to prevent hypoxemia and tissue hypoxia during the intubation procedure. For a patient breathing ambient air (i.e., room air), only 21% of the gas in the functional residual capacity is oxygen; 78% is nitrogen. Administering 100% oxygen to a patient prior to induction of anesthesia and tracheal intubation, referred to as "preoxygenation," can replace the nitrogen in the lung with oxygen, increasing up to five-fold the reservoir of oxygen available to the body during the procedure and prolonging the period during which intubation can be performed safely without encountering hypoxemia. In current clinical practice, the two most common methods of providing preoxygenation are:

1. Non-invasive positive pressure ventilation - a tight-fitting mask connected to either an invasive ventilator or non-invasive mechanical ventilator.
2. Facemask oxygen - with either a non-rebreather mask or a bag-mask device.

PREOXYGENATION WITH NON-INVASIVE POSITIVE PRESSURE VENTILATION:

Preoxygenation with non-invasive positive pressure ventilation is common during emergency tracheal intubation of critically ill adults in current clinical practice. During preoxygenation with non-invasive positive pressure ventilation, a tight-fitting mask is connected to a machine capable of providing positive pressure ventilation. Non-invasive positive pressure ventilation delivers up to 95-100% oxygen and can be provided by either a conventional invasive mechanical ventilator or a dedicated non-invasive ventilation machine, commonly referred to as a Bilevel Positive Airway Pressure (BiPAP) machine. In addition to providing high concentrations of oxygen, non-invasive positive pressure ventilation increases mean airway pressure and delivers breaths at a set rate during the period of hypopnea/apnea after induction. Because a mechanical ventilator is always required following intubation of a critically ill adult, no specialized equipment is required to use non-invasive positive pressure ventilation for preoxygenation of critically ill adults undergoing tracheal intubation.

PREOXYGENATION WITH FACEMASK OXYGEN:

In current clinical practice, preoxygenation with facemask oxygen is commonly performed using one of the following two types of facemask: [1] a non-rebreather mask or [2] a bag-mask device. Both a types of facemask (a non-rebreather and a compressed bag-mask device) deliver supplemental oxygen without increasing airway pressures or providing assistance with ventilation.

* A non-rebreather mask is a type of facemask with a loose-fitting mask that sits over a patient's nose and mouth and is connected to an oxygen reservoir. It delivers at least 15 liters per minute of 100% oxygen, but it may not reliably deliver flows of oxygen greater than 15 liters per minute and may allow entrainment of ambient air. Studies show that the while the oxygen content for healthy and calm volunteers may approach 100%, the oxygen content received by critically ill patients with tachypnea may be as low as 50%. It does not provide positive pressure.
* A bag mask device is a type of facemask with a mask that forms a tight seal over the mouth and nose when held in place by the operator, an exhalation port, and a self-inflating bag that serves as a reservoir for oxygen and can be compressed to provide positive pressure ventilation. If the bag of this device is compressed, this device delivers oxygen without providing positive pressure ventilation and can deliver more than 90% oxygen with an ideal mask seal. However, in the setting of emergency intubation leaks may result in the entrainment of ambient air and reduced oxygen delivery.

POTENTIAL ADVANTAGES OF PREOXYGENATION WITH NON-INVASIVE POSITIVE PRESSURE VENTILATION OR PREOXYGENATION WITH FACEMASK OXYGEN:

Preoxygenation with non-invasive positive pressure ventilation has been proposed to offer the following potential advantages compared to preoxygenation with facemask oxygen:

* Entrainment of ambient air: The tight-fitting mask used to deliver non-invasive ventilation entrains less ambient air than a non-rebreather or bag-mask device. The higher flow rates of oxygen gas with non-invasive ventilation may also help prevent entrainment of ambient air and increase the fraction of inspired oxygen.
* Atelectasis and alveolar recruitment: Preoxygenation and induction of anesthesia rapidly results in the development of atelectasis in both healthy patients and critically ill patients. This atelectasis increases shunt fraction and increases the risk of peri-procedural hypoxia. By delivering positive pressure during both inspiration and expiration, non-invasive ventilation raises mean airway pressure, recruiting alveoli and preventing the development of atelectasis.
* Hypopnea and Apnea. Administration of sedation and neuromuscular blocking agents reduces or eliminates spontaneous respiratory effort. This hypoventilation leads to accumulation of alveolar carbon dioxide and reductions in alveolar oxygen, contributing to hypoxemia. Use of non-invasive ventilation before induction and between induction and laryngoscopy provides continuous oxygen to the alveoli, increases the size of breaths taken in the setting of hypopnea, and delivers controlled breaths when patients are apneic.

Preoxygenation with facemask oxygen (via a non-rebreather or compressed bag-mask device) has been proposed to offer the following potential advantages compared with preoxygenation with non-invasive positive pressure ventilation:

* Simplicity of use: Preoxygenation with facemask oxygen (using either a non-rebreather or compressed bag-mask device) is simpler to set up than non-invasive positive pressure ventilation.
* Low risk of gastric insufflation: Although no clinical evidence exist to suggest that preoxygenation with non-invasive positive pressure ventilation increases the risk of gastric insufflation or aspiration of gastric contents, use of facemask oxygen (without any positive pressure) avoids this hypothetical concern.

PRIOR EVIDENCE FROM CLINICAL TRIALS:

Two small clinical trials have compared preoxygenation with non-invasive ventilation to preoxygenation with facemask oxygen during the tracheal intubation of critically ill adults. The first trial compared non-invasive ventilation to a facemask among 53 critically ill ICU patients in two hospitals and found that non-invasive ventilation increased the lowest oxygen saturation (93% vs. 81%, p<0.001) with no difference in incidence of aspiration (6% vs. 8%). The second trial compared non-invasive ventilation to a facemask oxygen with regard to severity of illness in the 7 days after intubation among 201 critically ill ICU patients. This trial found no significant difference in the severity of illness between groups and no significant difference in the rate of severe hypoxemia (18.4% vs 27.7%, p=0.10). This trial did not have adequate statistical power to detect clinically important differences between groups in the risk of hypoxemia. No large, multicenter trials have compared preoxygenation with non-invasive positive pressure ventilation to preoxygenation with facemask oxygen for critically ill adults undergoing tracheal intubation. Based on the available data from these small randomized clinical trials, preoxygenation with non-invasive positive pressure ventilation and preoxygenation with facemask oxygen both represent acceptable approaches to emergency tracheal intubation. Both approaches are considered standard-of-care and are used commonly in current clinical practice.

RATIONALE FOR A LARGE MULTICENTER TRIAL OF PREOXYGENATION:

Because of the imperative to optimize emergency tracheal intubation in clinical care, the common use of both preoxygenation with non-invasive positive pressure ventilation and preoxygenation with facemask oxygen in current clinical practice, and the lack of existing data from randomized trials to definitively inform whether preoxygenation strategy effects the rate of hypoxemia, examining the approach to preoxygenation during emergency tracheal intubation represents an urgent research priority. To address this knowledge gap, the investigators propose to conduct a large, multicenter, randomized clinical trial comparing preoxygenation with non-invasive positive pressure ventilation versus preoxygenation with facemask oxygen with regard to hypoxemic during tracheal intubation of critically ill adults in the ED or ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patient is located in a participating unit
* Planned procedure is tracheal intubation using a laryngoscope and sedation
* Planned operator is a clinician expected to routinely perform tracheal intubation in the participating unit.

Exclusion Criteria:

* Patient is receiving positive pressure ventilation by a mechanical ventilator, bag-mask device, or laryngeal mask airway
* Patient is known to be less than 18 years old
* Patient is known to be pregnant
* Patient is known to be a prisoner
* Immediate need for tracheal intubation precludes safe performance of study procedures
* Patient is apneic, hypopneic, or has another condition requiring positive pressure ventilation between enrollment and induction
* Operator has determined that preoxygenation with non-invasive positive pressure ventilation or preoxygenation with a facemask is required or contraindicated for optimal care of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1301 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-10-14 (Actual); Study Completion 2023-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Casey, MD, MSc, Principal Investigator — Vanderbilt University Medical Center; Adit A Ginde, MD, MPH, Principal Investigator — University of Colorado, Denver; Matthew W Semler, MD, MSc, Study Director — Vanderbilt University Medical Center; Kevin W Gibbs, MD, Study Chair — Wake Forest University Health Sciences
Locations (16):
- United States (16):
  - UAB Hospital, Birmingham, Alabama
  - University of Colorado Denver, Aurora, Colorado
  - University of Iowa, Iowa City, Iowa
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Ochsner Medical Center | Ochsner Health System, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor Scott & White Health, Temple, Texas
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Following publication, individual patient data will be made available for sharing to researchers with 1) a signed data access agreement, 2) research testing a hypothesis, 3) a protocol that has been approved by an institutional review board, and 4) a proposal that has received approval from the principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: Following publication. No end date
Access Criteria: 1. a signed data access agreement
  2. research testing a hypothesis
  3. a protocol that has been approved by an institutional review board
  4. a proposal that has received approval from the principal investigator

REFERENCES:
- [Derived] Gibbs KW, Semler MW, Driver BE, Seitz KP, Stempek SB, Taylor C, Resnick-Ault D, White HD, Gandotra S, Doerschug KC, Mohamed A, Prekker ME, Khan A, Gaillard JP, Andrea L, Aggarwal NR, Brainard JC, Barnett LH, Halliday SJ, Blinder V, Dagan A, Whitson MR, Schauer SG, Walker JE Jr, Barker AB, Palakshappa JA, Muhs A, Wozniak JM, Kramer PJ, Withers C, Ghamande SA, Russell DW, Schwartz A, Moskowitz A, Hansen SJ, Allada G, Goranson JK, Fein DG, Sottile PD, Kelly N, Alwood SM, Long MT, Malhotra R, Shapiro NI, Page DB, Long BJ, Thomas CB, Trent SA, Janz DR, Rice TW, Self WH, Bebarta VS, Lloyd BD, Rhoads J, Womack K, Imhoff B, Ginde AA, Casey JD; PREOXI Investigators and the Pragmatic Critical Care Research Group. Noninvasive Ventilation for Preoxygenation during Emergency Intubation. N Engl J Med. 2024 Jun 20;390(23):2165-2177. doi: 10.1056/NEJMoa2313680. Epub 2024 Jun 13. PMID 38869091
- [Derived] Gibbs KW, Ginde AA, Prekker ME, Seitz KP, Stempek SB, Taylor C, Gandotra S, White H, Resnick-Ault D, Khan A, Mohmed A, Brainard JC, Fein DG, Aggarwal NR, Whitson MR, Halliday SJ, Gaillard JP, Blinder V, Driver BE, Palakshappa JA, Lloyd BD, Wozniak JM, Exline MC, Russell DW, Ghamande S, Withers C, Hubel KA, Moskowitz A, Bastman J, Andrea L, Sottile PD, Page DB, Long MT, Goranson JK, Malhotra R, Long BJ, Schauer SG, Connor A, Anderson E, Maestas K, Rhoads JP, Womack K, Imhoff B, Janz DR, Trent SA, Self WH, Rice TW, Semler MW, Casey JD. Protocol and statistical analysis plan for the PREOXI trial of preoxygenation with noninvasive ventilation vs oxygen mask. medRxiv [Preprint]. 2023 Mar 24:2023.03.23.23287539. doi: 10.1101/2023.03.23.23287539. PMID 36993496

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Started | 645 | 656
Completed | 645 | 656
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group | Total
Number analyzed (Participants) | 645 | 656 | 1301
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [47 to 71] | 61 [47 to 70] | 61 [47 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 255 | 260 | 515
  Male | 390 | 396 | 786
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 384 | 399 | 783
  Non-Hispanic Black | 124 | 152 | 276
  Hispanic | 80 | 63 | 143
  Other | 48 | 36 | 84
  Not Reported | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 645 | 656 | 1301

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hypoxemia
Description: A peripheral oxygen saturation < 85% during the interval between induction and 2 minutes after tracheal intubation
Time Frame: from induction to 2 minutes following tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 624 | 637
Participants | 57 | 118

2. Secondary Outcome: Lowest Oxygen Saturation
Description: Lowest oxygen saturation during the interval between induction and 2 minutes after tracheal intubation
Time Frame: from induction to 2 minutes following tracheal intubation
Measure: Median (Inter-Quartile Range); unit: Oxygen Saturation (%)
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 624 | 637
Oxygen Saturation (%) | 99 [95 to 100] | 97 [89 to 100]

3. Other Pre Specified Outcome: Incidence of Operator-reported Aspiration
Time Frame: from induction to 2 minutes following tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 645 | 656
Participants | 6 | 9

4. Other Pre Specified Outcome: Fraction of Inspired Oxygen at 24 Hours After Induction
Time Frame: 24 hours after induction
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 590 | 594
Percentage | 40 [30 to 40] | 40 [30 to 40]

5. Other Pre Specified Outcome: Oxygen Saturation at 24 Hours After Induction
Time Frame: 24 hours after induction
Measure: Median (Inter-Quartile Range); unit: Oxygen Saturation (%)
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 589 | 594
Oxygen Saturation (%) | 97 [95 to 100] | 97 [95 to 100]

6. Other Pre Specified Outcome: Incidence of Pneumothorax
Description: Radiology report of new pneumothorax on chest x-ray in the 24 hours after induction
Time Frame: from induction to 24 hours after induction
Measure: Count of Participants; unit: Participants
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 509 | 497
Participants | 7 | 7

7. Other Pre Specified Outcome: Incidence of New Infiltrate
Description: Radiology report of new infiltrate on chest imaging in the 24 hours after intubation
Time Frame: from induction to 24 hours after induction
Measure: Count of Participants; unit: Participants
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 509 | 497
Participants | 144 | 148

8. Other Pre Specified Outcome: Incidence of Severe Hypoxemia
Description: Lowest oxygen saturation of <80% between induction and two minutes after tracheal intubation
Time Frame: from induction to 2 minutes following tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 624 | 637
Participants | 39 | 84

9. Other Pre Specified Outcome: Incidence of Very Severe Hypoxemia
Description: Lowest oxygen saturation of <70% between induction and two minutes after tracheal intubation
Time Frame: from induction to 2 minutes following tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 624 | 637
Participants | 15 | 36

10. Other Pre Specified Outcome: Oxygen Saturation at Induction
Time Frame: from enrollment to induction
Measure: Median (Inter-Quartile Range); unit: Oxygen Saturation (%)
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 625 | 643
Oxygen Saturation (%) | 100 [99 to 100] | 100 [97 to 100]

11. Other Pre Specified Outcome: Systolic Blood Pressure at Induction
Time Frame: from enrollment to induction
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 619 | 632
mmHg | 124 [107 to 143] | 129 [111 to 148]

12. Other Pre Specified Outcome: Duration From Induction to Successful Intubation
Time Frame: Duration of procedure (minutes)
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 645 | 656
Seconds | 115 [89 to 150] | 113 [85 to 152]

13. Other Pre Specified Outcome: Cormack-Lehane Grade of Glottic View on First Attempt
Description: Grade 1: Full view of glottis Grade 2: Partial view of glottis Grade 3: Only epiglottis seen (none of glottis) Grade 4: Neither glottis nor epiglottis seen
Time Frame: Duration of procedure (minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 645 | 655
Participants
  Grade 1 | 434 | 456
  Grade 2 | 165 | 148
  Grade 3 | 29 | 36
  Grade 4 | 17 | 15

14. Other Pre Specified Outcome: Incidence of Successful Intubation on the First Attempt
Description: Placement of an endotracheal tube in the trachea with a single insertion of a laryngoscope blade into the mouth and either a single insertion of an endotracheal tube into the mouth or a single insertion of a bougie into the mouth followed by a single insertion of an endotracheal tube into the mouth
Time Frame: Duration of procedure (minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 645 | 656
Participants | 534 | 535

15. Other Pre Specified Outcome: Number of Laryngoscopy Attempts
Time Frame: Duration of procedure (minutes)
Measure: Median (Inter-Quartile Range); unit: attempts
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 641 | 654
attempts | 1 [1 to 1] | 1 [1 to 1]

16. Other Pre Specified Outcome: Number of Attempts at Passing a Bougie
Time Frame: Duration of procedure (minutes)
Measure: Median (Inter-Quartile Range); unit: attempts
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 641 | 655
attempts | 0 [0 to 1] | 0 [0 to 1]

17. Other Pre Specified Outcome: Number of Attempts at Passing an Endotracheal Tube
Time Frame: Duration of procedure (minutes)
Measure: Median (Inter-Quartile Range); unit: attempts
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 641 | 654
attempts | 1 [1 to 1] | 1 [1 to 1]

18. Other Pre Specified Outcome: Incidence of Cardiovascular Collapse
Description: A composite of one or more of the following between induction and 2 minutes after intubation:
  * Systolic blood pressure < 65 mmHg
  * New or increased vasopressor
  * Cardiac arrest not resulting in death within 1 hour of induction
  * Cardiac arrest resulting in death within 1 hour of induction
Time Frame: from induction to 2 minutes following tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 645 | 656
Participants | 113 | 127

19. Other Pre Specified Outcome: 28-day In-hospital Mortality
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 645 | 656
Participants | 209 | 217

20. Other Pre Specified Outcome: Ventilator-free Days to 28 Days
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 645 | 656
Days | 21 [0 to 26] | 17 [0 to 25]

21. Other Pre Specified Outcome: ICU-free Days to 28 Days
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
Number analyzed (Participants) | 645 | 656
Days | 16 [0 to 23] | 14 [0 to 23]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to 28 days after enrollment.
Description: Because this trial compared strategies commonly used in routine clinical care, the only events that were recorded or reported as adverse events were those that were related to the study and serious or unexpected. Critically ill adults who require tracheal intubation are at risk for hypoxemia, hypotension, cardiac arrest, and death. These events were recorded as study outcomes and only recorded as AEs if related to the study intervention, which was expected to be rare.
Arm/Group | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group | Preoxygenation With Facemask Oxygen Group
All-Cause Mortality (participants affected / at risk) | 209/645 | 217/656
Serious Adverse Events (participants affected / at risk) | 2/645 | 0/656
Other Adverse Events (participants affected / at risk) | 0/645 | 0/656
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preoxygenation With Non-Invasive Positive Pressure Ventilation Group (N=645) | Preoxygenation With Facemask Oxygen Group (N=656)
Aspiration (Surgical and medical procedures) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT05267652/Prot_SAP_000.pdf